CLINICAL TRIAL: NCT07283744
Title: Project FIERCE - Fostering Internal and External Respect, Compassion, and Equanimity: A Mindfulness-Based Intervention to Reduce Stress Through the Cultivation of Loving-Kindness, Compassion, Joy, and Equanimity in Healthcare Professionals
Brief Title: A Mindfulness-Based Intervention to Reduce Stress Through the Cultivation of Loving-Kindness, Compassion, Joy, and Equanimity in Healthcare Professionals
Acronym: FIERCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Julienne Bower, PhD, Area Chair: Health Psychology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-25-1518
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Stress (Psychology); Inflamation; Psychosocial Functioning
Keywords: mindfulness; compassion; loving-kindness; healthcare professional; stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kindness and compassion-based meditation program (Experimental): Half of the participants will be randomly assigned to participate in the meditation intervention. This class will meet virtually once a week for six consecutive weeks, for one hour.
  Interventions: Behavioral: Building Emotional Strength Training
- Waitlist control (No Intervention): Half of the participants will be randomly assigned to the waitlist control. Participants assigned to this condition will have the opportunity to attend the meditation course after data collection is complete.

INTERVENTIONS:
Behavioral: Building Emotional Strength Training — The BEST intervention was designed as a secularized version of the traditional Four Immeasurables practice to promote the distinct emotional states of loving-kindness, compassion, sympathetic joy, and equanimity. Each session provides structured training and exercises in mindfulness, including formal meditation practices and strategies for the daily informal use of mindfulness, as well as opportunity for questions and group discussion. Home practice is a key component of BEST and is particularly important for addressing stress in daily life. Participants will be instructed to practice mindfulness techniques on a daily basis, beginning with five minutes and increasing to 20 minutes, with practice prior to work or other stress-inducing situations.
  Arms: Kindness and compassion-based meditation program

SUMMARY:
Nearly 50% of the adult workforce experience adverse psychological symptoms (e.g., stress, depression, burnout, etc.) stemming from workplace stressors, with healthcare workers experiencing rates as high as 80%. Some common complaints and downstream consequences of working in high-stress healthcare occupations are elevated levels of perceived stress, depression, and burnout. These conditions have been associated with unfavorable occupational (e.g., increased medical errors), patient (e.g., increased mortality rates), and provider-related outcomes (e.g., increased rates of cardiovascular disease), imposing a heavy burden on an already stretched system. Given the impact of perceived stress, depression, and burnout on employee and patient health, a clear need exists to develop effective interventions to reduce distress and promote well-being among healthcare professionals. In particular, interventions that target processes particularly vulnerable to provider stress (e.g., compassion) are needed.

The present study will evaluate the feasibility and efficacy of a mindfulness-based intervention inspired by the Buddhist Four Immeasurables practice on reducing perceived stress (primary outcome), depressive symptoms, burnout, and biological markers of inflammation, and enhancing psychological well-being and sleep quality (secondary outcomes) in 80 healthcare workers. Additionally, we will investigate several mediators (compassion, positive emotions, equanimity, and mindfulness) of intervention effects. Participants will be healthcare employees of UCLA Health. They will be enrolled in a six-week, two-arm randomized controlled trial. Participants will complete self-report questionnaires at baseline, mid-course, and post-intervention to assess study outcomes and mediators. We aim to advance the study of interventions that reduce distress and promote well-being using practices that cultivate kind feelings toward oneself and others.

DETAILED DESCRIPTION:
Healthcare providers face a large number of stressful situations daily, which may increase their risk of developing several adverse mental and physical health conditions. Some of the most common complaints and downstream consequences of working in high-stress healthcare occupations are elevated levels of perceptions of stress, depression, and burnout. Each of these conditions has been associated with a host of unfavorable occupational outcomes, including absenteeism, lost work productivity, increased medical errors, and poorer patient quality of care. Additionally, perceived stress, depression, and burnout have been associated with adverse provider outcomes, including increased rates of suicidality, substance misuse, exhaustion, musculoskeletal pain, and gastrointestinal complaints. Finally, these conditions impose a significant financial burden on an already strained healthcare system in the form of worker turnover and medical malpractice.

Overview: This single-site, two-arm, parallel-group RCT is designed to evaluate the feasibility and efficacy of a meditation-based intervention (Building Emotional Strength Training [BEST]) for perceived stress relative to a waitlist control for full-time healthcare workers. The intervention will be delivered by an experienced mediation instructor, following a manualized protocol, in a live online group format once a week for six consecutive weeks, held on Zoom. Groups will be conducted during the workday at standardized times. Assessments will be conducted both before and after the intervention to evaluate the effects of the intervention on the outcome.

Participants: Study participants will be 80 full-time healthcare workers employed by UCLA Health. They will be recruited in cohorts of 20-30 and randomized 1:1 to one of the two study arms. Participants will complete questionnaires and undergo blood collection on their own, which will be conducted before and after the six-week intervention. Additionally, several mechanisms of intervention effects will be assessed at the midpoint of the intervention (week three of the six-week intervention). Following CONSORT guidelines, we have designated one primary outcome for this trial: perceived stress. Additional (secondary) outcomes include symptoms of burnout, depression, subjective sleep quality, psychological well-being, and inflammatory processes, all of which have been associated with healthcare provider health and well-being and have been shown to be sensitive to the effects of meditation interventions. Further, several theory-based mechanisms of intervention effects include self-compassion, compassion for others, positive and negative emotions, equanimity, and mindfulness, all of which are plausible pathways through which meditation-based interventions may influence perceived stress.

Eligibility Screening, Enrollment, and Baseline Assessment (T1). Potential participants will be directed to contact the study coordinator via email or phone. Research staff will then contact potential participants by phone to confirm eligibility criteria. The 4-item Perceived Stress Scale will be used to screen for at least moderate levels of stress. Those who score a "5" or above, indicating at least moderate levels of stress, will be considered eligible for study participation. Participants will be recruited in cohorts of 20-30 healthcare providers, who will be randomly assigned to either the BEST group or the waitlist control, allowing for our desired mindfulness group size of 10-15 participants. Screening will continue until we have an adequate number of eligible, interested, and available participants for the next cohort.

All participants who are determined to be eligible will then review and verbally acknowledge the IRB-approved consent form. After obtaining consent and enrollment, participants will be emailed a link to complete the study questionnaires. The questionnaires will include the following: Background demographic and medical characteristics, health behaviors, Perceived Stress Scale (PSS), Maslach Burnout Inventor for Medical Personnel (MBI-M), Center for Epidemiological Studies-Depression (CES-D), Mental Health Continuum Short Form (MHC-SF), Insomnia Severity Index (ISI), Self-Compassion Scale (SCS), Compassion Scale (CS), modified Differential Emotions Scale (mDES), Equanimity Scale (ES), Five Factor Mindfulness Questionnaire (FFMQ).

They will also receive an at-home blood collection kit in the mail to provide a blood sample for immune evaluation. Participants will provide blood samples for immune evaluation using the Tasso OnDemand device, which allows self-collection of a single capillary blood sample and does not require venipuncture. The Tasso device sticks to the skin with a light adhesive. When the button is pressed, a vacuum forms and a lancet pricks the surface of the skin. The vacuum draws blood out of the capillaries and into a sample pod attached to the bottom of the device. Participants will watch a demonstration video during their baseline assessment visit, and then use the device to collect a blood sample. Approximately 1/8th of a teaspoon of blood will be drawn at each in-person assessment. Participants will be advised to complete the blood collection in the morning to control for diurnal variations in immune parameters.

Baseline assessments will be conducted during the 2 weeks preceding the onset of intervention. Study staff completing the eligibility screening, consent, and emailing participants the assessment links will be blind to participant group assignment.

Randomization. Upon completion of the baseline assessment, participants will be randomized 1:1 to one of the two study conditions using the Qualtrics randomization feature by the study coordinator. The randomization feature on Qualtrics will be used to randomize participants. The study coordinator will inform participants of their assigned condition and provide them with information on the intervention (e.g., class dates and times, Zoom link, etc.).

Interventions: The intervention will be delivered remotely via Zoom. Group sessions will be conducted during the workday (around lunchtime).

Building Emotional Strength Training (BEST). The experimental mindfulness intervention was designed as a secularized version of the traditional Four Immeasurables practice. Diana Winston, Director of UCLA Mindful, developed the intervention based on her decades of experience working with new meditation practitioners and her expertise in designing group-based mindfulness courses for various audiences. In particular, she adapted a class previously offered through the Mindful Awareness Research Center (MARC) that focused on positive affect. Notably, the research team consulted with several healthcare professionals at UCLA to determine the most suitable delivery format, intervention duration, and optimal time of day for holding the intervention classes.

The traditional Four Immeasurables practice includes exercises to promote the distinct emotional states of loving-kindness, compassion, sympathetic joy, and equanimity. The BEST curriculum is a six-week, group-based program where participants attend one class per week for six consecutive weeks. Each session focuses on a different component of the Four Immeasurables practice. During the one-hour class, participants will receive structured training and instruction in mindfulness exercises. The instructor will provide theoretical information and formal instructions on practicing the day's specific topic and will allow students to ask questions to enhance their learning.

Additionally, participants will be guided through each meditation exercise introduced during class. Furthermore, each class will include dyadic discussions, allowing participants to interact directly with one another. The sessions will introduce the following topics and associated practices: 1) introduction to mindfulness, 2) further development of mindfulness, 3) loving-kindness, 4) compassion, 5) joy, and 6) equanimity.

The BEST intervention also includes home practice, in which participants are encouraged to practice the meditation technique introduced in class that week at home, starting with five minutes and gradually increasing to 20 minutes per day throughout the six weeks of the intervention. Diana Winston will teach all classes.

Waitlist Control (WLC). The WLC will control for naturally occurring changes in the outcomes and mediators over the assessment period. Participants in this group will not engage in any study-related activities outside of the remote assessments. Participants randomized to this condition will be offered the BEST intervention after all data collection is completed.

Mid-Course Assessment (T2). At the halfway point of the intervention, all participants will be emailed a link to complete self-report questionnaires assessing the primary outcome and mediator variables only.

Post-Intervention Assessment (T3). All participants will be emailed the post-intervention assessment link and mailed a second blood collection kit to complete both tasks within 2 weeks following the conclusion of the study intervention. The questionnaire will include all study variables.

ELIGIBILITY:
Inclusion Criteria: 1) full-time physician (M.D. or D.O.), 2) at least 18 years of age, 3) able to attend the six-week intervention, 4) fluent in English, and 5) access to the internet and email.

Exclusion Criteria. 1) having a current and consistent meditation practice (i.e., engaging in a formal meditation practice at least three days per week for five minutes each day), 2) previous participation in a Four Immeasurable course (e.g., attending a Brahmaviharas meditation retreat), 3) absence of at least mild levels of perceived stress as determined by a score less than five on the four-item Perceived Stress Scale (PSS-4; 92), 4) regular tobacco use (given its impact on immune function; 90), and 5) failure to agree to the informed consent. The presence or absence of perceived stress will be assessed using the PSS-4 during the initial phone screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Perceived Stress as Assessed by the Perceived Stress Scale | At baseline, mid-course at week 3, and post-intervention at week 6.
  Stress will be assessed using the ten-item Perceived Stress Scale (PSS). The PSS evaluates how often individuals appraised situations in their lives as stressful during the past month (e.g., "In the last month, how often have you been angered because of things that were outside of your control?"). Respondents respond on a five-point Likert scale from 0 (never) to 4 (very often). All scores are summed to provide a total stress score. Scores range from 0 to 40, with higher scores indicating a higher level of perceived stress. The PSS has been widely used with healthcare professional populations and has been shown to be responsive to mindfulness-based interventions.

SECONDARY OUTCOMES:
Mean Change from Baseline in Depressive Symptoms as Assessed with the Center for Epidemiological Studies Depression Scale | At baseline and post-intervention at week 6.
  Depressive symptoms will be based on scores on the 20-item Center for Epidemiologic Studies-Depression Scale (CES-D), a commonly used depression measure. The CES-D is a reliable, validated, and widely used measure that includes central components of depressive symptomatology, including depressed mood, worthlessness, hopelessness, loss of appetite, and psychomotor retardation. Respondents respond to twenty statements that assess how often the individual felt or behaved during the past week (e.g., "I felt that I could not shake off the blues even with help from my family and friends") on a four-point Likert scale from 0 (rarely or none of the time [less than 1 day]) to 3 (most or all of the time [5-7 days]). All 20 items will be summed to provide a total score. The possible range of scores is 0-60, with higher scores indicating a greater frequency of depressive symptoms. The CES-D has frequently been used to assess depressive symptoms in healthcare workers.
Mean Change from Baseline in Burnout as Assessed with the Maslach Burnout Inventory for Medical Personnel | At baseline and post-intervention at week 6.
  Burnout will be measured via the 22-item Maslach Burnout Inventory for Medical Personnel (MBI-M). The MBI-M measures three components of burnout: emotional exhaustion, depersonalization, and reduced personal accomplishment. Emotional exhaustion refers to feeling emotionally overextended and exhausted by one's work. Depersonalization refers to an impersonal response toward the recipients of one's services. Personal accomplishment refers to feelings of competence and achievement in work-related pursuits. Items are scored on a 7-point Likert scale from 0 (never) to 6 (every day). Higher scores on the emotional exhaustion and depersonalization subscales correspond to a greater experience of burnout. The personal accomplishment subscale is positively worded; therefore, a one-item increase corresponds to a greater experience of work-related efficacy. Each subscale will be summed, providing a total score for emotional exhaustion, depersonalization, and personal accomplishment.
Mean Change from Baseline in Psychological Well-being as Assessed with the Mental Health Continuum Short Form | At baseline and post-intervention at week 6.
  Well-being will be measured using the 14-item Mental Health Continuum Short Form (MHC-SF). The MHC-SF is a 14-item scale that measures three dimensions of psychological well-being: hedonic, eudaimonic-social, and eudaimonic-psychological. Hedonic well-being refers to pleasurable states characterized by the presence of positive and absence of negative affect. Eudaimonic social well-being refers to flourishing within a social context characterized by social coherence and actualization. Eudaimonic psychological well-being refers to a sense of living a life of purpose, characterized by feelings of personal growth and self-actualization. Respondents respond to the fourteen items to assess how often they felt concerning the statements during the past month, using a six-point Likert scale ranging from 0 (never) to 5 (every day). All scores are summed to provide a total well-being score. The possible range of scores is 0-70, with higher scores indicating greater subjective well-being.
Mean Change from Baseline in Sleep Quality as Assessed with the Insomnia Severity Index | At baseline and post-intervention at week 6.
  Sleep quality will be assessed using the seven-item Insomnia Severity Index (ISI). The ISI is a reliable and valid self-report measure that evaluates the severity and impact of insomnia over the past two weeks. Respondents are asked to respond to the seven items to assess how they relate to each statement over the past two weeks, using a five-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores are summed to obtain a total score. The possible range of scores on the ISI is 0-28, with higher scores indicating more severe insomnia. Additionally, scores of 15 or higher are indicative of clinically significant insomnia. The ISI has been validated for use with healthcare professionals and shown to be responsive to mindfulness interventions.
Mean Change from Baseline in Inflammation as Assessed by Circulating IL-6, IL-8, IL-10, TNF-alpha, and IFN-gamma and Molecular Analysis of Gene Expression and Signaling of 19 Pro-Inflammatory, 28 Type I Interferon Response, and 3 Antibody Synthesis Genes | At baseline and post-intervention at week 6.
  We will utilize an integrated assessment of inflammation that encompasses systemic levels of inflammatory markers, inflammatory gene expression, and promoter-based bioinformatics analyses of specific inflammation-related transcription factors. Each measurement level provides unique and complementary information, offering a comprehensive view of inflammatory activity.

OTHER OUTCOMES:
Mean Change from Baseline in Self-compassion as Assessed with the Self-Compassion Scale | At baseline, mid-course at week 3, and post-intervention at week 6.
  Self-compassion will be assessed using the 12-item Self-Compassion Scale-Short Form (SCS-SF). The SCS-SF assesses an individual's global tendency to show kindness, concern, and sympathy for one's own suffering. The scale has six subscales with two items each: self-kindness (compassion for oneself during difficult moments), self-judgment (disapproval or intolerance of oneself), common humanity (appreciation of the universal nature of having flaws and inadequacies), isolation (experiencing failures alone), mindfulness (balance and poise during difficult moments), and over-identification (obsessing over negative feelings). Individuals answer how often they generally behave in a stated manner on a five-point Likert scale from 1 (almost never) to 5 (almost always) in response to the 12 items. Scores range from 1 - 5, with higher scores indicating greater feelings of self-compassion. The SCS-SF has been used in the context of an intervention for healthcare workers.
Mean Change from Baseline in Compassion for Others as Assessed with the Compassion Scale | At baseline, mid-course at week 3, and post-intervention at week 6.
  Compassion for others will be assessed using the 16-item Compassion Scale (CS) (129). The CS comprises four subscales, each with four items, that determine how one generally reacts toward others. The four subscales include kindness (compassion and caring towards others during times of difficulty), common humanity (appreciation for the universal experience of pain), mindfulness (awareness of others and their experiences), and indifference (an unsympathetic demeanor towards the suffering of others). Individuals answer how often they generally behave in a stated manner on a five-point Likert scale from 1 (almost never) to 5 (almost always) in response to the 16 items. The mean of each subscale is then calculated to compute a total mean (the average of the six subscale means). Scores range from 1 - 5, with higher scores indicating greater feelings of compassion for others. The CS has been used in healthcare worker populations .
Mean Change from Baseline in Positive and Negative Emotions as Assessed with the modified Differential Emotions Scale | At baseline, mid-course at week 3, and post-intervention at week 6.
  Positive emotions will be assessed using the 20-item modified Differential Emotions Scale (mDES) (133). The mDES is based on Fredrickson's Broaden-and-Build theory of positive emotions and assesses the degree to which individuals experience a spectrum of discrete positive and negative emotions within a given timeframe. The questionnaire includes ten items assessing positive emotions, such as contentment, amusement, and awe, and ten items assessing negative emotions, such as sadness, shame, anger, and hatred. The mDES attempts to capture the experience of both high and low arousal positive and negative emotions. For each item, respondents indicate the extent to which they felt a specific emotion in the past 24 hours on a five-point Likert scale, ranging from 0 (not at all) to 4 (extremely). Each subscale (positive and negative) is independent of the other, so the mDES will yield a total score for both positive and negative emotions. Scores on each subscale range from 0 to 40.
Mean Change from Baseline in Equanimity as Assessed with the Equanimity Scale | At baseline, mid-course at week 3, and post-intervention at week 6.
  Equanimity will be assessed using the 16-item Equanimity Scale (ES-16). The ES-16 assesses the tendency of an individual to act in a balanced, calm, and even-tempered manner toward all experiences (positive or negative). The scale comprises two subscales, each consisting of eight items: experiential acceptance (neutrality toward all internal experiences) and non-reactivity (an evenness of response toward all experiences). Example items include, "When I experience distressing thoughts and images, I can accept the experience," and "I can pay attention to what is happening in my body without disliking or wanting more of the feeling or sensation." Individuals respond on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) to indicate how they view themselves. The eight items from the non-reactivity subscale are reverse-scored. All 16 items are summed to provide a total score. Scores range from 16 - 80, with higher scores indicating greater levels of equanimity.
Mean Change from Baseline in Mindfulness as Assessed with the Five Factor Mindfulness Questionnaire | At baseline, mid-course at week 3, and post-intervention at week 6.
  Mindfulness will be assessed using the 15-item Five Factor Mindfulness Questionnaire (FFMQ-15). The FFMQ assesses five distinct facets of mindfulness using five subscales: observing (e.g., "I pay attention to how my emotions affect my thoughts and behavior"), describing (e.g., "I can usually describe how I feel at the moment in considerable detail"), acting with awareness (reverse scored; e.g., "I am easily distracted"), non-judging (reverse scored; e.g., "I criticize myself for having irrational or inappropriate emotions"), and non-reactivity ("I perceive my feelings and emotions without having to react to them"). Individuals respond on a five-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true), to indicate how each statement relates to their general attitude. All items are summed and divided by 15 to provide an average mindfulness score. Scores range from 1 - 5, with higher scores indicating greater mindfulness.
Acceptability of the BEST Intervention as Assessed with the Treatment Satisfaction Questionnaire | Post-intervention at week 6.
  The acceptability of the intervention will be evaluated using an abbreviated and adapted version of the Treatment Satisfaction Questionnaire (TSQ), administered at the post-intervention assessment (T3). The three-item TSQ determines the extent to which the participant views the intervention as helpful and beneficial. Respondents respond to three statements assessing their agreement and general perception of the intervention on an eight-point Likert scale, ranging from 0 (not at all) to 7 (extremely). Example items include "The intervention was useful for me" and "The intervention improved my quality of life." All three items are summed to provide a total satisfaction score. The possible range of scores is 0-21, with higher scores indicating greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julienne E Bower, Ph.D., Principal Investigator — University of California, Los Angeles, Psychology Department
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any individual participant data (IPD) with any other researchers. Data will be reported in group form to prevent personal identification of participants. When the research has been completed, the data will be stored in a secured area of a private, locked research office. Any personal identifiers and/or codes linking the data to personal identifiers will be kept on a separate computer with password protection for reference and for future research. All personal identifiers will be kept confidential. Only identified members of the research team and the P.I. will have access to the data, identifiers and/or codes. Data with subject identifiers will not be released to any agency or persons.